CLINICAL TRIAL: NCT01021085
Title: Evaluation Of A Fetal Sex Determination Test At 36-56 Days Gestation In Assisted Reproductive Technology (ART) Achieved Pregnancies
Brief Title: Evaluation of Fetal Sex in Assisted Reproductive Technology (ART) Achieved Pregnancies
Acronym: PREVIEW
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SQNM-IVF-FS-102
Record Dates: First submitted 2009-10-29; First posted 2009-11-26 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Fetal Sex Determination
Keywords: Assisted Reproductive Technology; circulating cell free fetal DNA; First trimester

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Maternal whole blood and urine will be collected. Whole blood will be processed to plasma and buffy coat.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women who have conceived via ART and are between days 36 and 56 of gestation

SUMMARY:
Whole blood and urine samples will be collected from pregnant woman of gestational age 36-56 days as confirmed by artificial reproductive technology (ART). The samples will be used to develop a prenatal sex test using circulating cell free fetal DNA (ccffDNA) in maternal plasma or urine.

DETAILED DESCRIPTION:
This is an observational study whereby samples will be tested to determine the presence or absence of fetal Y chromosome genes to test for the fetal sex of the baby. The blood draw and urine collection will occur between 36-42, 43-49, and 50-56 days gestation. The fetal gender will be requested at or soon after delivery. The accuracy of the test and the optimal time to perform the test during pregnancy will be assessed by comparing the test results from maternal blood and/or urine samples obtained between days 36 and 56 of gestation to the fetal sex results obtained at birth.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-45 years of age inclusive
* Subject is female
* Subject is pregnant
* Gestational age can be determined via IVF or IUI
* Subject is 36-42 days pregnant as determined by IVF transfer or IUI
* Subject agrees to provide 3 separate blood and urine samples

Exclusion Criteria:

* None

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who are pregnant via assisted reproductive technology between days 36 and 56 gestational age
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-04; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Develop a prenatal sex test using blood and/or urine samples from pregnant women. | 36 to 56 days of gestation

SECONDARY OUTCOMES:
Establish the earliest time point between days 36 and 56 of gestation that the prenatal sex test has optimal performance. | 36 to 56 days of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Allan Bombard, MD MBA, Study Director — Sequenom, Inc.
Locations (3):
- United States (3):
  - San Diego Fertility Center, San Diego, California
  - Fertility Centers of Illinois, Glenview, Illinois
  - Fertility Center of Las Vegas, Las Vegas, Nevada